CLINICAL TRIAL: NCT04710589
Title: Clinical Target Volume Exploration of 3D Printing Personalized Template Assisted CT-guided Radioactive Iodine-125 Seeds Implantation as a Salvage Treatment for Recurrent Rectal Cancer Patients After Operation and Radiotherapy
Brief Title: CTV Exploration of 3D-PT Assisted CT-guided I-125 Seeds Implantation for Recurrent Rectal Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CTV of 125I for rectal cancer
Record Dates: First submitted 2020-12-30; First posted 2021-01-14 (Actual); Last update posted 2021-01-14 (Actual); Status verified 2021-01

CONDITIONS: Recurrent Rectal Cancer; 125I Seeds Implantation; Clinical Target Volume
Keywords: recurrent rectal cancer; 125I seeds implantation; clinical target volume; 3D printing template; radiotherapy
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CTV 3mm: CTV is expanded by 3mm on the basis of GTV.
- CTV 6mm: CTV is expanded by 6mm on the basis of GTV.
  Interventions: Radiation: CTV

INTERVENTIONS:
Radiation: CTV — According to the clinical conditions of the patients, they will be assigned to two groups based on the doctor's recommendations and their own wishes
  Groups: CTV 6mm

SUMMARY:
This study is to explore the progression-free survival time (PFS) , overall survival time (OS), quality of life and side effects between two different clinical target volumes in the treatment of 3D printing template-assisted CT-guided radioactive iodine-125 seeds implantation for recurrent rectal cancer after surgery and radiotherapy and investigate the clinical and dosimetric prognosis factors for outcomes.

DETAILED DESCRIPTION:
From June 2019 to December 2020 in each participating center, patients with recurrent rectal cancer after surgery and radiotherapy will be included in the study if they meet the inclusion criteria and do not meet the exclusion criteria. According to the clinical conditions of the patients, they will be assigned to groups A or B according to the doctor's recommendations and their own wishes. GTV of both groups are visible tumors. The CTV of group A is expanded by 3mm on the basis of GTV, and the CTV of group B is expanded by 6mm. Both groups A and B received prescription dose: 95% GTV (120-160) Gy, 95% CTV (90-120) Gy. The activities of 125I seeds will be 0.4mCi-0.7mCi. All patients will receive 3D printed template-assisted 125I seeds implantation and be followed up. The differences in local progression-free survival time, overall survival time, change of quality of life, and side effects between different groups will be prospectively analyzed.

ELIGIBILITY:
Inclusion Criteria:

* KPS score above 60;
* Age from 18 to 80 years old;
* Rectal cancer by histological diagnosis, recurrence after surgery and radiotherapy;
* The diameter of the lesion ≤ 5cm;
* The tumor has not invaded the intestines or bladder;
* The estimated survival time is more than 3 months;
* The percutaneous puncture path is feasible and the preoperative plan can meet the prescription dose;
* Blood routine, liver, kidney and other major organ functions: WBC is normal, PLT≥100×109/L, HGB≥100g/L; urea nitrogen, creatinine≤1.25×upper limit of normal (UNL), ALT (SGPT) and AST (SGOT) ≤2.5×UNL; ECG is basically normal;
* Recurrence in pelvic region after surgery and radiotherapy for various reasons; or oligo-metastatic lesions less than 3, which are stable with treatment. Except for rectal incision stump and recurrence at the anastomosis.

Exclusion Criteria:

* Major organ failure, decompensated heart and lung failure such as congestive heart failure, coronary heart disease with clinical symptoms, and arrhythmia that cannot be controlled by drugs;
* Patients with other serious uncontrollable medical diseases;
* Severe coagulation dysfunction;
* With serious infection or ulcer at the puncture site;
* Pregnancy, breastfeeding women, children and mental patients;
* Patients with severe diabetes;
* Cases that invade large blood vessels and vital organs, which may cause hemorrhage and severe organ dysfunction;
* Those who have participated in clinical trials of other drugs or medical devices before being selected but have not reached the time limit of the main research endpoint or have completed clinical trials of other drugs or medical devices for less than 4 weeks;
* Poor compliance and unable to complete the course of treatment;
* Other reasons the researchers think it is inappropriate to participate in this clinical trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Recurrent rectal cancer after surgery and radiotherapy who will receive 3D-PT Assisted CT-guided I-125 Seeds Implantation
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression free survival time (PFS) | 3 years
  The time from 125I radioactive seeds implantation to local failure or death.

SECONDARY OUTCOMES:
Overall survival time (OS) | 3 years
  The time from 125I radioactive seeds implantation to death due to any cause.

OTHER OUTCOMES:
Karnosky Score | 3 years
  This is a functional status score, which is one of the methods to evaluate the quality of life. The range is from 0-100 points. The higher the score, the better the functional status and the higher the quality of life are.
Visual Analogue Score | 3 years
  This is a pain score ,which is one of the evaluation indicators of quality of life. The range is 0-10 points. The higher the score, the higher the pain and the worse the quality of life are.
Side effects | 3 years
  Difined and classified by RTOG

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Unnversity Third Hospital, Beijing, Beijing Municipality, China